CLINICAL TRIAL: NCT03477526
Title: Status and Develepment Mental Quality of Life in Lung Fibrosis in Comparison of COPD Inpatients Before and After Pulmonary Rehabilitation
Brief Title: Status and Develepment Mental Quality of Life COPD/IPF Inpatients Before and After Pulmonary Rehabilitation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PhD Student stopped working on this project
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: Lungenfibrose e.V. (Unknown)
Responsible Party: Principal Investigator, Klaus Kenn, Principal Investigator, Schön Klinik Berchtesgadener Land
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Fibrosis 2016
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Idiopathic Pulmonary Fibrosis and COPD
Keywords: pulmonary fibrosis; COPD; pulmonary rehabilitation; mental status (anxiety and depression); quality of life; physical activity
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Disease, Chronic Obstructive; Pulmonary Fibrosis; Anxiety Disorders; Depression; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD patients (GOLD stage III-IV) (Experimental)
  Interventions: Procedure: Pulmonary rehabilitation program
- IPF patients (Active Comparator)
  Interventions: Procedure: Pulmonary rehabilitation program

INTERVENTIONS:
Procedure: Pulmonary rehabilitation program — 3 weeks, ...

SUMMARY:
As the result of our last study "Long Term effects of an Inpatient Pulmonary Program in Patients with Pulmonary Fibrosis" already demonstrated the positive effects of a Pulmonary Rehabiliation on the mental status. In this current study the aim will be to analyse the personality type regarding anxiety and depression

ELIGIBILITY:
Inclusion Criteria:

* COPD GOLD III-IV
* IPF according Pulmonary Guidelines

Exclusion Criteria:

< 30% FVC comorbidities with a negativ influence on the prognosis neurological and orthopaedic deficits, which make the participation of the pulmonary rehabilitation impossible non-compliance no written informed consent of the patient

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Anxiety score | 3 weeks
  Hospital Anxiety and Depression scale

SECONDARY OUTCOMES:
Anxiety score | 3 months
  Hospital Anxiety and Depression scale

CONTACTS AND LOCATIONS:
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Germany

IPD SHARING:
Plan to Share IPD: Undecided